CLINICAL TRIAL: NCT01614392
Title: Lower Extremity Muscle and Function in the Elderly: Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Roger A Fielding, Director and Senior Scientist, Professor of Nutrition, Jean Mayer USDA Human Nutrition Research Center on Aging., Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG-18844
Record Dates: First submitted 2009-09-28; First posted 2012-06-07 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Mobility Limitation
Keywords: Resistance Exercise; Physical Activity; Mobility disability; Physical function; Muscle Strength; Older Adults; Mobility-Limited; Peak power and strength
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High velocity low force Power Training (Experimental): Lower Extremity high velocity power training performed at lower external resistance (40% of the 1 repetition maximum muscle strength). Leg and knee extension exercises were performed twice per week (3 sets of each exercise consisting of 10 repetitions).
  Interventions: Behavioral: High velocity low force Power Training
- Low velocity high force Power Training (Experimental): Lower extremity low velocity power training performed at high external resistance (70% of the 1 repetition maximum muscle strength). Leg and knee extension exercises were performed twice per week (3 sets of each exercise consisting of 10 repetitions).
  Interventions: Behavioral: Low velocity high force Power Training

INTERVENTIONS:
Behavioral: High velocity low force Power Training — Lower Extremity high velocity power training performed at lower external resistance (40% of the 1 repetition maximum muscle strength). Leg and knee extension exercises were performed twice per week (3 sets of each exercise consisting of 10 repetitions).
  Arms: High velocity low force Power Training
Behavioral: Low velocity high force Power Training — Lower extremity low velocity power training performed at high external resistance (70% of the 1 repetition maximum muscle strength). Leg and knee extension exercises were performed twice per week (3 sets of each exercise consisting of 10 repetitions).
  Arms: Low velocity high force Power Training

SUMMARY:
This research study is looking to compare the effects of two uniquely different power training interventions (high force, lower velocity versus low force, high velocity) on changes in mobility status among older individuals at risk for mobility disability.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female 70-85 yrs
* Community dwelling
* Short Performance Battery Score >9
* BMI range 19-32 kg/m2
* Willingness to be randomized and come the laboratory for 20 weeks.

Exclusion Criteria:

* Acute or Terminal Illness
* MI in previous 6 months, symptomatic coronary artery disease or congestive heart failure.
* Upper or Lower extremity fracture in previous 6 months
* Uncontrolled hypertension (150/90mmHg)
* Neuromuscular diseases and drugs that affect neuromuscular function
* Hormone replacement therapy
* Participation in any regular endurance or resistance training exercise during previous 3 months

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Fieilding, Ph D., Principal Investigator — Jean Mayer USDA Human Nutrition Research Center on Aging
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Velocity Low Force Power Training | Low Velocity High Force Power Training
Started | 25 | 27
Completed | 24 | 24
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Velocity Low Force Power Training | Low Velocity High Force Power Training | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.3 (5) | 77.6 (4) | 77.9 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Leg Extensor Muscle Power
Description: Leg extensor muscle power measured on pneumatic strength testing equipment at a external force consistent with 70% of the participant maximum leg extensor strength.
Time Frame: Change from baseline to Week 16
Population: 4 participants dropped out of study before follow up
Measure: Mean (Standard Error); unit: Watts
Groups:
- Power Training Performed at Low External Resistance: High velocity low force power training performed at low external resistance (40% of the 1repetition maximum strength (RM)[LO]
- Power Training Performed at High External Resistance: Low velocity high force power training performed at high external resistance (70% of the 1 repetition maximum (RM) [HI])
Arm/Group | Power Training Performed at Low External Resistance | Power Training Performed at High External Resistance
Number analyzed (Participants) | 24 | 24
Watts | 32.9 (13) | 41.6 (12)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | High Velocity Low Force Power Training | Low Velocity High Force Power Training
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 1/25 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Velocity Low Force Power Training (N=25) | Low Velocity High Force Power Training (N=27)
General (Infections and infestations) | 1 | 3 — Upper respiratory infection
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 1 — Hamstring and back pain
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Exacerbation of COPD
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 1 — Non-injurious fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No